CLINICAL TRIAL: NCT05638503
Title: Multi-center Study on New Cardiovascular Remodeling and Function Parameters in Hypertension
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: QLCR20220272
Record Dates: First submitted 2022-11-15; First posted 2022-12-06 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
Keywords: Hypertension; Echocardiography; Cardiovascular remodeling
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertension with left ventricular hypertrophy group: 2015 ASE/EACVI guideline standard: Eccentric hypertrophy, EH: LVMI>115g/ m2（male）or LVMI>95g/ m2（female）and RWT≤0.42 Concentric hypertrophy, CH: LVMI>115g/ m2（male）or LVMI>95g/ m2（female）and RWT>0.42
  Reference Values for Chinese (EMINCA) and Configuration Analysis Based on Ganau Typing:
  Eccentric hypertrophy, EH: LVMI>108g/ m2（male）and RWT≤0.51or LVMI>99g/ m2（female）and RWT≤0.49 Concentric hypertrophy, CH: LVMI>108g/ m2（male）and RWT>0.51 or LVMI>99g/ m2（female）and RWT>0.49
  Interventions: Other: Left ventricular hypertrophy
- Hypertension with left ventricular non-hypertrophy group: 2015 ASE/EACVI guideline standard: Normal left ventricular geometry, NG: LVMI≤115g/m2（male）or LVMI≤95g/m2（female）and RWT≤0.42 Concentric remodeling, CR: LVMI≤115g/m2（male）or LVMI≤95g/ m2（female）and RWT>0.42
  Reference Values for Chinese (EMINCA) and Configuration Analysis Based on Ganau Typing:
  Normal left ventricular geometry, NG: LVMI≤108g/ m2（male）and RWT≤0.51 or LVMI≤99g/ m2（female）and RWT>0.49 Concentric remodeling, CR: LVMI≤108g/ m2（male）and RWT>0.51 or LVMI≤99g/ m2（female）and RWT>0.49
  Interventions: Other: Left ventricular non-hypertrophy

INTERVENTIONS:
Other: Left ventricular hypertrophy — Hypertension with normal left ventricular geometry and left ventricular concentric remodeling
  Groups: Hypertension with left ventricular hypertrophy group
Other: Left ventricular non-hypertrophy — Hypertension with left ventricular concentric hypertrophy and left ventricular eccentric hypertrophy
  Groups: Hypertension with left ventricular non-hypertrophy group

SUMMARY:
The investigators want to explore the relationship between different configurations of hypertension and the incidence of cardiovascular events by the guidelines reference range and EMINCA recommended reference range. Then the investigators want to enroll twenty research centers and 2200 hypertensions were planned to be collected and followed up in the 12th, 24th, 36th and 48th months after being enrolled in this study. Physical examination, ECG examination, laboratory examination, echocardiography and carotid ultrasound should be taken when baseline and follow-up. Echocardiographic measurement parameters were analyzed and the relationship between the echocardiographic measurement parameters and cardiovascular events and prognosis of hypertension.

DETAILED DESCRIPTION:
Different configurations of hypertension are important risk factor for the morbidity and mortality of cardiovascular and cerebrovascular diseases in China. Studies have shown that left ventricular hypertrophy (LVH) and left atrial enlargement caused by hypertension are independent risk factors for cardiovascular events. The LVM and LAV derived from the normal value data of Chinese healthy adults have been reported to be different from the recommended reference values in guidelines, and the distribution characteristics of hypertension remodeling are also different. However, the characteristics and outcomes of cardiac remodeling in Chinese hypertensive population and whether this difference in configuration has an impact on the treatment, prognosis and cardiovascular events of hypertensive population are still needed to be explored.

This study was to observe the relationship between blood pressure and cardiovascular remodeling evaluated by different standards in hypertensive population, and compare the relationship between different cardiac configurations and cardiovascular events in Chinese hypertensive population.

Twenty research centers and 2200 hypertensions were planned to be collected and followed up in the 12th, 24th, 36th and 48th months after being enrolled in this study. Physical examination, ECG examination, laboratory examination, echocardiography and carotid ultrasound should be taken when baseline and follow-up.

Echocardiographic measurement parameters including M-mode and two-dimensional ultrasonic parameters; doppler ultrasound parameters; relevant parameters of two-dimensional speckle tracking, myocardial work parameters; the left ventricular remodeling parameters (LVM and RWT); cardiac morphological changes; three-dimensional ultrasound parameters were analyzed and the relationship between the echocardiographic measurement parameters and cardiovascular events and prognosis of hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-75 years old;
2. No antihypertensive drugs were used and three blood pressure measurements were conducted on different days, with systolic blood pressure ≥ 140 mmHg (1 mmHg=0.133 kPa) and/or diastolic blood pressure ≥ 90 mmHg; or have a history of hypertension and are using antihypertensive drugs, even if the blood pressure is lower than 140/90 mmHg;
3. Left ventricular ejection fraction was normal (LVEF ≥ 0.5).
4. All patients agreed to participate in the experiment and signed the informed consent form.

Exclusion Criteria:

1. Secondary hypertension caused by renal parenchymal diseases, renal vascular diseases, coarctation of aorta and endocrine system diseases;
2. Severe cardiovascular and cerebrovascular diseases; heart valve disease; persistent atrial fibrillation and severe arrhythmia; previously undergone cardiovascular disease surgery;
3. Abnormal liver function; abnormal renal function and diabetes;
4. Pregnant or breastfeeding women;
5. Expected survival time due to non-cardiovascular disease<4 years;
6. Patients with poor echocardiographic image quality.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No antihypertensive drugs were used and three blood pressure measurements were conducted on different days, with systolic blood pressure ≥ 140 mmHg (1 mmHg=0.133 kPa) and/or diastolic blood pressure ≥ 90 mmHg; or have a history of hypertension and are using antihypertensive drugs, even if the blood pressure is lower than 140/90 mmHg
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Emerging atrial fibrillation | Through study completion, on average once a year.
  The differences in the incidence of atrial fibrillation between the two groups
Emerging unstable angina, myocardial infarction, heart failure, coronary revascularization, cardiovascular death | Through study completion, on average once a year.
  The differences in the incidence of unstable angina, myocardial infarction, heart failure, coronary revascularization, cardiovascular death between the two groups
Emerging transient ischemic attack (TIA) or stroke | Through study completion, on average once a year.
  The differences in the incidence of transient ischemic attack (TIA) or stroke between the two groups

SECONDARY OUTCOMES:
Emerging decreased cardiac function with preserved ejection fraction | Through study completion, on average once a year.
  The differences between the two groups in the incidence of decreased cardiac function with preserved ejection fraction measured by echocardiography compared to that at the baseline
Emerging cardiac remodeling | Through study completion, on average once a year.
  The differences between the two groups in the incidence of cardiac remodeling measured by echocardiography compared to that at the baseline
Emerging aortic aneurysm or aortic dissection | Through study completion, on average once a year.
  The differences in the incidence of aortic aneurysm or aortic dissection between the two groups
Emerging serious arrhythmias | Through study completion, on average once a year.
  ECG showed that QTc (QT interval corrected by heart rate) was more than 500ms or QTc was longer than the baseline level for more than 60ms, emerging torsade de pointes ventricular tachycardia and other serious arrhythmias
The relationship between the deviations of blood pressure within the same day and the difference of cardiac function indexes | Through study completion, on average once a year.
  The differences between the two groups in the incidence of the deviations between blood pressure and cardiac function parameters at the same day measured by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Mei Zhang, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-08-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT05638503/Prot_000.pdf
  • Informed Consent Form (2022-08-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT05638503/ICF_001.pdf